CLINICAL TRIAL: NCT04561297
Title: Assessing the Utility of Tissue Dielectric Constant (TDC) Measurements to Differentiate Breast Cancer From Healthy Breasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Surgical Specialists of Miami (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-7-Non-NSU Health
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: tissue dielectric constant; breast cancer; tumor; biopsy
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients scheduled for biopsy of the breast
Masking Description: Measurements are made prior to the biopsy determination of whether tumor is benign or malignant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Biopsied Patients (Experimental): Patients scheduled for a breast biopsy will have breast tissue dielectric constant measurements made prior to the biopsy
  Interventions: Diagnostic Test: TDC differential value

INTERVENTIONS:
Diagnostic Test: TDC differential value — TDC measurements in all patients agreeing to participate who are scheduled for a biopsy of a breast tumor or mass

SUMMARY:
Patients with pending breast biopsies will have the tumor site's tissue dielectric constant (TDC) measured prior to the biopsy. Similar TDC measurements will be made at a standard breast site on the biopsied breast and on mirrored sites on the non-affected breast.

DETAILED DESCRIPTION:
Patients with pending breast biopsies will have the tumor site's tissue dielectric constant (TDC) measured prior to the biopsy. Similar TDC measurements will be made at a standard breast site on the biopsied breast and on mirrored sites on the non-affected breast. Values obtained at the biopsy site will be compared against the outcome of the biopsy analysis: benign vs. malignant. In addition the measurements obtained at the standardized site for all breasts will be used to establish a set of reference values to characterize breast TDC values. In addition, inter-breast differentials will be used to characterize these ranges for future studies and clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* You must be scheduled for a breast biopsy of a breast mass or abnormality with the collaborating centers

Exclusion Criteria:

* You have any open wounds over the breasts
* You have had breast cancer
* You have or have had breast implants or have undergone any breast surgery or breast biopsy
* You have any implantable wires, this includes a Pacemaker, Implantable Cardioverter ° Defibrillators (ICDs), and/or Left Ventricular Assist Device (LVAD)
* You are pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be scheduled for a breast biopsy with the collaborating centers
Enrollment: 60 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
TDC Tumor Differential | one hour
  Difference between TDC values measured at tumor site between benign vs. malignant
TDC Inter-Breast Differentials | one hour
  Difference between TDC values measured at corresponding sites betweenbreasts
TDC reference values for breasts | one hour
  Composite reference ranges for TDC values as measured on standard breast site of all

CONTACTS AND LOCATIONS:
Locations (1):
- Surgical Specialists of Miami, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No